CLINICAL TRIAL: NCT03229655
Title: Evaluation of Sequential Stent Addition vs. Incremental Dilation & Stent Exchange for Management of Anastomotic Biliary Strictures After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: University of Rochester (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Division of Gastroenterology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41606
Record Dates: First submitted 2017-06-30; First posted 2017-07-25 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Anastomotic Stenosis; Biliary Stricture
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential stent addition (Experimental): ERCP with sphincterotomy and stent placement is initially performed, then additional stents are placed across the stricture during sequential ERCPs, without stent removal/exchange or stricture dilation.
  Interventions: Procedure: Protocol for increasing number of stents across the anastomosis
- Incremental Dilation & Stent Exchange (Active Comparator): ERCP with sphincterotomy and stent placement is initially performed, with subsequent ERCPs involving removal of previously placed stents, stricture dilation and balloon sweeps to extract stone debris/sludge.
  Interventions: Procedure: Protocol for increasing number of stents across the anastomosis

INTERVENTIONS:
Procedure: Protocol for increasing number of stents across the anastomosis — Sequential placement of straight plastic biliary stents across the duct-to-duct anastomosis without dilation or stent exchange. Multiple ERCPs will be performed with addition of a single stent at each ERCP until the final ERCP when all stents will be removed.

SUMMARY:
Prospective, randomized comparison of the incremental dilation and stent exchange vs. sequential stent addition approaches for management of anastomotic biliary strictures will facilitate optimal management of patients who develop anastomotic biliary strictures after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Clinical concern for anastomotic biliary stricture following liver transplantation (as determined by the referring transplant hepatologist)
3. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Age <18
2. Potentially vulnerable subjects including, homeless people, pregnant females, employees and students.
3. Complex post-surgical anatomy e.g. Choledochojejunostomy, Billroth type II anatomy, Roux-en-Y-gastrojejunostomy
4. Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
5. Other biliary process which accounts for patient's abnormal liver function studies/imaging (i.e. significant non-anastomotic biliary stricture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic biliary stricture resolution | Immediately following final ERCP with stent removal
  Fluoroscopic (on ERCP image) resolution of stricture at the time of final study ERCP when all stents are removed

SECONDARY OUTCOMES:
Fluoroscopy Parameters | 1 day
  Fluoroscopy Time per fluoroscopy machine output
Adverse Events | 1 week
  Pancreatitis, bleeding, infection, perforation to be assessed one day and one week post-procedure
Sustained resolution of anastomotic stricture for 6 months | 6 months after final study ERCP with stent removal
  No evidence of recurrent stricture based on clinical status and laboratory studies
Sustained resolution of anastomotic stricture for 12 months | 12 months after final study ERCP with stent removal
  No evidence of recurrent stricture based on clinical status and laboratory studies

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No